CLINICAL TRIAL: NCT02976519
Title: A Phase Ib, Multicentre, Double Blind, Randomized, Two-part Study, First Part Multiple Rising Dose and Second Part Two-way Cross-over, to Assess Safety, Tolerability, Efficacy and Pharmacokinetics of BI 443651 Compared to Placebo Via Respimat® in Healthy Volunteers and CF Subjects.
Brief Title: BI 443651 Multiple Rising Dose in Healthy Volunteers Followed by a Cross-over in CF Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1363.2; 2016-001504-31 (EudraCT Number)
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 443651 (Experimental)
  Interventions: Drug: BI 443651
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 443651 — twice daily
  Arms: BI 443651
Drug: Placebo — twice daily
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the safety, tolerability, and pharmacokinetics of BI 443651 in male and female healthy volunteers and subjects with Cystic Fibrosis (CF).

ELIGIBILITY:
Inclusion criteria:

Healthy volunteers:

* Signed informed consent
* Healthy male or female subjects
* - Women of childbearing potential (WOCBP) should only be dosed after a confirmed menstrual period and/or with a progesterone level at Day -5 to Day -3 that demonstrates a dip from baseline, indicating a menstrual bleed prior to dosing.
* Age of 18 to 55 years (incl.)
* Body mass index (BMI) of 18.5 to 32.0 kg/m2 (incl.)
* Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) of equal or greater than 80% of predicted normal, at screening and prior to randomisation

Cystic Fibrosis (Cross over part):

* Signed informed consent
* Males or females with a documented diagnosis of cystic fibrosis
* Women of childbearing potential (WOCBP) should only be dosed after a confirmed menstrual period and/or with a progesterone level at Day -5 to Day -3, that demonstrates a dip from baseline, indicating a menstrual bleed prior to dosing. For CF subjects of child bearing potential this must confirmed prior to second treatment period.
* Age 18 to 55 years (each inclusive)
* BMI of 18 to 32.0 kg/m2 (incl.)
* Pre-bronchodilator FEV1 >/= to 70% of predicted normal at screening and prior to randomisation
* Clinical stability as defined by no evidence of acute upper or lower respiratory tract infection; no pulmonary exacerbation requiring use of i.v. / oral / inhaled antibiotics, or oral corticosteroids; no change in pulmonary disease therapy; if on cycling antibiotics, these must be initiated within 2 weeks prior to randomisation; no acute (serious or non-serious) illness not related to cystic fibrosis; no infection with an organism associated with more rapid decline in pulmonary function (eg, Burkholderia cenocepacia, B dolosa, or Mycobacterium abscessus).
* Able to perform technically acceptable pulmonary functions test (PFTs)
* Further inclusion criteria apply.

Exclusion criteria:

* Any evidence of a concomitant disease judged as clinically relevant by the investigator including gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, dermatologic, hematologic, neurological and psychiatric, oncological, coagulation or hormonal disorders as determined by medical history, examination, and clinical investigations at screening that may, in the opinion of the investigator, result in any of the following:

  * Put the subject at risk because of participation in the study.
  * Influence the results of the study.
  * Cast doubt on the subject's ability to participate in the study.
* Chronic or relevant acute infections.
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* History of myocardial infarction; history of acute coronary syndrome
* History of and/or active life-threatening cardiac arrhythmia, as assessed by the investigator
* Major surgery (major according to the investigator's assessment)
* History of chronic kidney disease (estimate glomerular filtration rate (EGFR) <59 mls/min including corrections as per ethnicity)
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Unsuitable veins for venipuncture (for instance, veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture) as assessed by the investigator
* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG) is deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, specifically volunteers with serum potassium > upper limit of normal should be excluded; Safety laboratory screening and Day -7 to Day -3, evaluation can be repeated twice during screening.
* For healthy volunteers, repeated measurement (i.e. > 2 measurements) of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg. Volunteers will be excluded with a pulse rate outside the range of 45 to 90 bpm.
* A marked baseline prolongation of mean QT/QTcF interval (such as QTcF intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening or prior to randomisation
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome).
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTcF interval
* Intake of drugs with a long half-life (more than 24hrs) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication unless this is allowed medications.
* CF subjects treated with non-permitted concomitant medication. Specifically medications causing changes in serum potassium are restricted
* Current or previous participation in another interventional trial, including where an investigational drug has been or will be administered within 60 days or 5 half-lives (whichever is longer) prior to screening
* For healthy volunteers and CF subjects: current smokers or ex-smokers of less than 12 months and/or with a pack year history of more than 5 years
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Lungenärztliche Praxis, München-Pasing
- United Kingdom (2):
  - Celerion Inc, Belfast
  - The Medicines Evaluation Unit, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 2 parts. The first part was a multiple rising dose (MRD) trial in healthy participants. The second part followed a cross-over design with respect to placebo and BI 443651 treatment in participants with cystic fibrosis. Both parts were randomised, placebo-controlled, and double-blinded.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that they (all participants) met all inclusion/exclusion criteria. Participants were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Placebo Matching BI 443651: Healthy participants were treated with placebo matching to BI 443651 via Respimat® inhaler twice daily for 6.5 days in Part 1.
- BI 443651 100 Microgram (μg): Healthy participants were treated with BI 443651 100 μg dose via Respimat® inhaler twice daily for 6.5 days in Part 1.
- BI 443651 400 μg: Healthy participants were treated with BI 443651 400 μg dose via Respimat® inhaler twice daily for 6.5 days in Part 1.
- BI 443651 1200 μg: Healthy participants were treated with BI 443651 1200 μg dose via Respimat® inhaler twice daily for 6.5 days in Part 1.
- BI 443651 1800 μg: Healthy participants were treated with BI 443651 1800 μg dose via Respimat® inhaler twice daily for 6.5 days in Part 1.
- BI 443651 600 μg/ Placebo Matching BI 443651: Participants suffering from cystic fibrosis were treated with 600 μg BI 443651 dose in period 1 and followed by placebo matching to BI 443651 in period 2, both administered via Respimat® inhaler twice daily for 13.5 days treatment periods separated by a wash-out period of at least 30 days between drug administrations in Part 2.
- Placebo Matching BI 443651/ BI 443651 600 μg: Participants suffering from cystic fibrosis were treated with placebo matching to BI 443651 in period 1 and followed by 600 μg BI 443651 dose in period 2, both administered via Respimat® inhaler twice daily for 13.5 days treatment periods separated by a wash-out period of at least 30 days between drug administrations in Part 2.
Period: Treatment Period 1 (Part 1 and Part 2)
Arm/Group | Placebo Matching BI 443651 | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg | BI 443651 600 μg/ Placebo Matching BI 443651 | Placebo Matching BI 443651/ BI 443651 600 μg
Started (Started are treated) | 8 | 8 | 8 | 8 | 8 | 12 | 12
Completed | 8 | 7 | 8 | 7 | 8 | 12 | 12
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Wash-out Period (Part 2 Only)
Arm/Group | Placebo Matching BI 443651 | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg | BI 443651 600 μg/ Placebo Matching BI 443651 | Placebo Matching BI 443651/ BI 443651 600 μg
Started | 0 | 0 | 0 | 0 | 0 | 12 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 12 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Reason not listed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2 (Part 2 Only)
Arm/Group | Placebo Matching BI 443651 | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg | BI 443651 600 μg/ Placebo Matching BI 443651 | Placebo Matching BI 443651/ BI 443651 600 μg
Started | 0 | 0 | 0 | 0 | 0 | 12 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 12 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all randomised subjects who had been treated with at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 443651 | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg | BI 443651 600 μg/ Placebo Matching BI 443651 | Placebo Matching BI 443651/ BI 443651 600 μg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (7.9) | 39.1 (10.2) | 38.9 (9.4) | 32.1 (8.1) | 41.1 (10.4) | 38.3 (12.4) | 34.0 (8.1) | 37.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 8
  Male | 8 | 8 | 8 | 8 | 8 | 9 | 7 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 5
  White | 7 | 6 | 7 | 5 | 8 | 12 | 11 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAE) Over the Treatment Period in Part 1 and Part 2
Description: Percentage of participants with treatment-emergent adverse events (TEAE) over the treatment period in Part 1 and Part 2. For Part 1: From the first dose of study medication up to 30 days after the day of last intake of study medication, up to 44 days. For Part 2: From the first dose of study medication up to 30 days after the day of last intake of study medication, up to 51 days.
Time Frame: Up to 44 days (for Part 1) or 51 days (for Part 2) (Please check the measure description for detailed timeframe)
Population: TS
Measure: Number; unit: Percentage of participants (%)
Groups:
- Placebo Matching BI 443651 600 μg: Participants suffering from cystic fibrosis were treated with placebo matching to BI 443651 600 μg dose via Respimat® twice daily for 13.5 days in Part 2.
- BI 443651 600 μg: Participants suffering from cystic fibrosis were treated with BI 443651 600 μg dose via Respimat® twice daily for 13.5 days in Part 2.
Arm/Group | Placebo Matching BI 443651 | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg | Placebo Matching BI 443651 600 μg | BI 443651 600 μg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 24 | 22
Percentage of participants (%) | 37.5 | 62.5 | 87.5 | 100.0 | 87.5 | 58.3 | 59.1

2. Secondary Outcome: Maximum Measured Concentration of the BI 443651 in Plasma After the Administration of the First Dose (Cmax) on Day 1 and Over the Time Interval From 0 to 12 h After the 13th Dose (Cmax,13) on Day 7, in Part 1
Description: Maximum measured concentration of the BI 443651 in plasma after the administration of the first dose (Cmax) on day 1 and over the time interval from 0 to 12 h after the 13th dose (Cmax,13) on day 7, in Part 1. Pharmacokinetic samples were collected at 00:15 hours:minutes (h:m) pre-dose and at 00:15, 00:30, 00:45, 1:00, 2:00, 4:00, 6:00, 8:00 and 11:45 h:m after first drug administration on day 1 (for Cmax) and after last drug administration on day 7 (for Cmax,13).
Time Frame: Day 1 and Day 7 (Please check the measure description for detailed timeframe)
Population: Pharmacokinetic (PK) set (PKS): The PKS included all subjects in the TS who provided at least 1 PK parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole (pmol)/Litre (L)
Arm/Group | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg
Number analyzed (Participants) | 8 | 7 | 8 | 8
picomole (pmol)/Litre (L)
  Cmax | 158 (60.8) | 782 (46.8) | 3400 (64.7) | 6320 (48.2)
  Cmax,13: number analyzed (Participants) | 7 | 7 | 7 | 8
  Cmax,13 | 250 (31.9) | 745 (70.3) | 4000 (27.2) | 6060 (70.6)
Statistical Analysis 1: Comparison: BI 443651 100 Microgram (μg) vs BI 443651 400 μg vs BI 443651 1200 μg vs BI 443651 1800 μg; Cmax. The basic model used for the investigation of dose proportionality was a power model (regression model applied to log-transformed data) that described the functional relationship between the dose and PK endpoints; Test type: Other; Slope = 1.2705, 95% CI 2-sided [1.1067 to 1.4343], Standard Error of Mean 0.0801 — Based on the estimate for slope parameter (β), a 2-sided 95% confidence interval (CI) for the slope was computed. Standard error of the mean is actually standard error of slope
Statistical Analysis 2: Comparison: BI 443651 100 Microgram (μg) vs BI 443651 400 μg vs BI 443651 1200 μg vs BI 443651 1800 μg; Cmax,13. The basic model used for the investigation of dose proportionality was a power model (regression model applied to log-transformed data) that described the functional relationship between the dose and PK endpoints; Test type: Other; Slope = 1.1361, 95% CI 2-sided [0.9598 to 1.3123], Standard Error of Mean 0.0859 — Based on the estimate for slope parameter (β), a 2-sided 95% CI for the slope was computed. Standard error of the mean is actually standard error of slope

3. Secondary Outcome: Area Under the Concentration-time Curve of the BI 443651 in Plasma Over the Time Interval From 0 to 12 Hours After the Administration of the First Dose (AUC0-12) on Day 1 and After the 13th Dose (AUC0-12,13) on Day 7 in Part 1
Description: Area under the concentration-time curve of the BI 443651 in plasma over the time interval from 0 to 12 hours (h) after the administration of the first dose (AUC0-12) on day 1 and after the 13th dose (AUC0-12,13) on day 7 in Part 1. Pharmacokinetic samples were collected at 00:15 h:m pre-dose and at 00:15, 00:30, 00:45, 1:00, 2:00, 4:00, 6:00, 8:00 and 11:45 h:m after first drug administration on day 1 (for AUC0-12) and after last drug administration on day 7 (for AUC0-12,13).
Time Frame: Day 1 and Day 7 (Please check the measure description for detailed timeframe)
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg
Number analyzed (Participants) | 8 | 7 | 8 | 8
pmol*h/L
  AUC0-12 | 409 (50.5) | 1980 (47.7) | 9150 (59.6) | 16200 (43.9)
  AUC0-12,13: number analyzed (Participants) | 7 | 7 | 7 | 8
  AUC0-12,13 | 868 (35.3) | 2260 (54.0) | 12200 (37.6) | 18400 (54.6)
Statistical Analysis 1: Comparison: BI 443651 100 Microgram (μg) vs BI 443651 400 μg vs BI 443651 1200 μg vs BI 443651 1800 μg; AUC0-12. The basic model used for the investigation of dose proportionality was a power model (regression model applied to log-transformed data) that described the functional relationship between the dose and PK endpoints; Test type: Other; Slope = 1.2743, 95% CI 2-sided [1.1231 to 1.4255], Standard Error of Mean 0.0739 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: BI 443651 100 Microgram (μg) vs BI 443651 400 μg vs BI 443651 1200 μg vs BI 443651 1800 μg; AUC0-12,13. The basic model used for the investigation of dose proportionality was a power model (regression model applied to log-transformed data) that described the functional relationship between the dose and PK endpoints; Test type: Other; Slope = 1.0924, 95% CI 2-sided [0.9296 to 1.2551], Standard Error of Mean 0.0793 — [estimate comment as in outcome 2, analysis 2]

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 30 days after the day of last intake of study medication, up to 37 days (for Part 1) and up to 44 days (for Part 2).
Description: Treated set (TS): The TS included all randomised subjects who had been treated with at least 1 dose of trial medication.
Arm/Group | Placebo Matching BI 443651 | BI 443651 100 Microgram (μg) | BI 443651 400 μg | BI 443651 1200 μg | BI 443651 1800 μg | Placebo Matching BI 443651 600 μg | BI 443651 600 μg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/8 | 0/8 | 0/8 | 1/24 | 0/22
Other Adverse Events (participants affected / at risk) | 3/8 | 5/8 | 7/8 | 8/8 | 7/8 | 8/24 | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 443651 (N=8) | BI 443651 100 Microgram (μg) (N=8) | BI 443651 400 μg (N=8) | BI 443651 1200 μg (N=8) | BI 443651 1800 μg (N=8) | Placebo Matching BI 443651 600 μg (N=24) | BI 443651 600 μg (N=22)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 443651 (N=8) | BI 443651 100 Microgram (μg) (N=8) | BI 443651 400 μg (N=8) | BI 443651 1200 μg (N=8) | BI 443651 1800 μg (N=8) | Placebo Matching BI 443651 600 μg (N=24) | BI 443651 600 μg (N=22)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 5 | 1 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 5 | 4 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 2 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 4 | 1 | 6 | 5
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medical device site rash (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT02976519/SAP_000.pdf
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02976519/Prot_001.pdf